CLINICAL TRIAL: NCT00000210
Title: Treatment Efficacy for Drug Abuse and AIDS Prevention
Brief Title: Treatment Efficacy for Drug Abuse and AIDS Prevention - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Mclean Hospital (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NIDA-06116-1; R18-06116-1
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2002-12

CONDITIONS: Cocaine-Related Disorders; Heroin Dependence
Keywords: opioid addiction; cocaine addiction
MeSH Terms: conditions — Cocaine-Related Disorders; Heroin Dependence; Opioid-Related Disorders | interventions — Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of buprenorphine for treatment of concurrent intravenous heroin and cocaine dependence.

ELIGIBILITY:
Please contact site for information.

Ages: 26 Years to 41 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1989-09; Primary Completion 1996-02 (Actual); Study Completion 1996-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack Mendelson, M.D., Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Dept. of Psychiatry, Belmont, Massachusetts, United States